CLINICAL TRIAL: NCT06548906
Title: A Trial Investigating the Pharmacokinetics, Pharmacodynamics and Safety of GZR4 Injection at Different Injection Regions in Healthy Subjects
Brief Title: A Study of GZR4 Injection at Different Injection Sites
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GZR4-T2D-103
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GZR4 Injection- Abdomen (Experimental): Participants received GZR4 Injection by subcutaneous injection on Abdomen.
  Interventions: Drug: GZR4 Injection
- GZR4 Injection- Upper Arm (Experimental): Participants received GZR4 Injection by subcutaneous injection on Upper Arm.
  Interventions: Drug: GZR4 Injection
- GZR4 Injection- Thigh (Experimental): Participants received GZR4 Injection by subcutaneous injection on Thigh.
  Interventions: Drug: GZR4 Injection

INTERVENTIONS:
Drug: GZR4 Injection — GZR4 Injection administered sc, once weekly.

SUMMARY:
This trial is conducted in China. This study is a randomized, single-center, open, three-period crossover trial in healthy subjects to compare the PK, PD, and safety of a single administration of GZR4 at different injection sites (abdomen, deltoid region of upper arm, and thigh).

ELIGIBILITY:
Inclusion Criteria:

* 1. Signing the informed consent form (ICF) before the trial, fully understanding the trial content, process and possible adverse reactions, and being able to comply with the contraindications and restrictions specified in this protocol.
* 2. A Male adult subjects aged 18-55 years old.
* 3. Body mass index (BMI) between 19.0-24.0 kg/m2

Exclusion Criteria:

* 1. Known or suspected hypersensitivity to investigational medical product(s) or related products.
* 2. Participation in a clinical study of another study drug within 3 months prior to randomization.
* 3. Physical examination, vital signs, laboratory examination, imaging examination, 12-lead electrocardiogram and other auxiliary examination results that the researchers considered abnormal clinical significance during screening.
* 4. Donation of blood or blood products (more than 100mL) or significant blood loss (more than 200 mL) within 6 months prior to screening
* 5. More than 14 units of alcohol per week within 3 months prior to randomization
* 6. Smoking more than 5 cigarettes per day within 3 months prior to randomization

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
AUC0-672h | From Predose to 672 hours after a single dose
  Area Under the Concentration Versus Time Curve of GZR4 Injection From Time Zero to 672 hours

SECONDARY OUTCOMES:
AUC0-∞ | From Predose to 672 hours after a single dose
  Area Under the Concentration Versus Time Curve of GZR4 Injection From Time Zero to Infinity
Cmax | From Predose to 672 hours after a single dose
  Maximum Concentration of GZR4 Injection

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Study Site, Beijing, China

IPD SHARING:
Plan to Share IPD: No